CLINICAL TRIAL: NCT03271567
Title: Detection of Circulating Mycobacterium Tuberculosis Antigen Peptides for the Diagnosis of Active Pulmonary and Extrapulmonary Tuberculosis in Hospitalized Patients
Brief Title: Nanodisk-MS Assay for the Diagnosis of Active Pulmonary and Extrapulmonary Tuberculosis in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Alice Ho Miu Ling Nethersole Hospital (Other)
Responsible Party: Principal Investigator, Grace Lui, Associate consultant, Chinese University of Hong Kong
Other Study IDs: TB Protocol ver.1
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Active Tuberculosis; Tuberculosis, Extrapulmonary; Tuberculosis, Pulmonary
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis, Extrapulmonary; Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nanodisk-MS assay — Nanodisk-MS assay is a recently reported novel assay for quantitative detection of various MTB antigen peptides, using nanotechnology and mass spectrometry that showed remarkable sensitivity and specificity in diagnosing active pulmonary and extrapulmonary TB. This assay detected MTB-specific antigens, CFP-10 and ESAT-6, in patients' serum samples.

SUMMARY:
Diagnosis and treatment of tuberculosis are often delayed in hospitalized patients, leading to worse outcomes. Rapid diagnosis of tuberculosis currently relies on microscopy and molecular techniques, which have limitations including low sensitivity and high cost.Highly sensitive diagnostic technique is needed for more accurate rapid diagnosis of tuberculosis to aid earlier initiation of antituberculous therapy. Detection of Mycobacterium tuberculosis (MTB) antigens in the bloodstream can potentially allow early diagnosis of tuberculosis. This study aims to evaluate the diagnostic performance of a novel assay using nanotechnology to detect MTB antigens in patients admitted to hospital with suspected pulmonary and/or extrapulmonary tuberculosis. Blood will be taken from eligible patients, and will be sent to the School of Biological and Health Systems Engineering, Arizona State University, for detection of 10-kDa culture filtrate protein (CFP-10) and the 6 kDa early secretory antigenic target (ESAT-6), two antigens specific for MTB, using the Nanodisk-MS assay. Investigations, including microscopy, culture, MTB polymerase chain reaction (PCR), and imaging, will be performed for diagnosis of tuberculosis. The diagnostic performance of Nanodisk-mass spectrometry (MS) assay will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 or above,
* Assessed by an Infectious Diseases physician to have clinical and/or radiological suspicion of pulmonary and/or extrapulmonary TB.

Exclusion Criteria:

* Refusal to consent from patients or next of kins for incompetent patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Prince of Wales Hospital and the Alice Ho Miu Ling Nethersole Hospital with suspected pulmonary and extrapulmonary TB will be identified by Infectious Diseases physician and recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic test correlation | One year from the date of recruitment
  Sensitivity, specificity, positive predictive value, and negative predictive value, will be calculated to determine accuracy of Nanodisk-MS assay, in diagnosing "culture-positive" and "culture-negative" pulmonary and/or extrapulmonary TB.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Yan Grace Lui, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Liu C, Zhao Z, Fan J, Lyon CJ, Wu HJ, Nedelkov D, Zelazny AM, Olivier KN, Cazares LH, Holland SM, Graviss EA, Hu Y. Quantification of circulating Mycobacterium tuberculosis antigen peptides allows rapid diagnosis of active disease and treatment monitoring. Proc Natl Acad Sci U S A. 2017 Apr 11;114(15):3969-3974. doi: 10.1073/pnas.1621360114. Epub 2017 Mar 27. PMID 28348223
- [Background] Lui G, Wong RY, Li F, Lee MK, Lai RW, Li TC, Kam JK, Lee N. High mortality in adults hospitalized for active tuberculosis in a low HIV prevalence setting. PLoS One. 2014 Mar 18;9(3):e92077. doi: 10.1371/journal.pone.0092077. eCollection 2014. PMID 24642794